CLINICAL TRIAL: NCT00897507
Title: Single Nucleotide Polymorphisms and Relapse Risk in Standard Risk ALL
Brief Title: DNA Analysis of Tumor Tissue Samples From Young Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL04B2; NCI-2009-00309 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000371580; COG-AALL04B2; AALL04B2; AALL04B2 (Other: Childrens Oncology Group); AALL04B2 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2017-10

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission; Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ancillary-Correlative (genotype assessment): Tumor tissue samples undergo genotype assessment on the Pyrosequencing platform. Contingency tables and X^2 test performs a univariate analysis of the risk of relapse and genotype, and multivariable analyses using logistic regression. Cox proportional hazards evaluate the risk of relapse given genotype and other confounders. Genotype patterning, classification and regression trees, and multifactor dimensionality reduction evaluates for patterns of single nucleotide polymorphisms associated with toxicity and relapse risk.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This laboratory study is looking at DNA in tumor tissue samples from young patients with acute lymphoblastic leukemia. DNA analysis of tumor tissue may help doctors predict how well patients will respond to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To validate significant associations between SNPs and treatment outcome and toxicity on Children's Cancer Group (CCG)-1891 on an independent sample set from a successor CCG study for standard risk acute lymphoblastic leukemia (ALL), CCG-1952.

II. To evaluate the role of SNPs in drug metabolizing enzymes and the development of veno-occlusive disease in patients on CCG-1952.

III. To evaluate interactions among genotypes and other risk factors for treatment response in a combined data set of CCG-1891 and CCG-1952 with recently developed analytic tools for high dimensional data.

IV. To develop predictive models utilizing genetic information obtained in Aim 1.1 and clinical data to predict treatment response and toxicity.

OUTLINE:

Tumor tissue samples undergo genotype assessment on the Pyrosequencing platform. Contingency tables and X^2 test performs a univariate analysis of the risk of relapse and genotype, and multivariable analyses using logistic regression. Cox proportional hazards evaluate the risk of relapse given genotype and other confounders. Genotype patterning, classification and regression trees, and multifactor dimensionality reduction evaluates for patterns of single nucleotide polymorphisms associated with toxicity and relapse risk.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in clinical trial CCG-1891 or CCG-1952 with pediatric ALL

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2004-05-13 (Actual); Primary Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Leukemia Relapse | Day 7
  Contingency tables will be used to tabulate the relationship between relapse and genotype, race, leukemia cytogenetics, day 7 bone marrow status, and treatment arm
Development of veno-occlusive disease in patients on CCG-1952 | Day 28
  Classification and Regression Trees (CART), genotype patterning, Multifactor Dimensionality Reduction (MDR) techniques will be used to identify SNP combinations associated with risk of relapse and VOD
Development of a predictive model of leukemia relapse | Day 28
  Predictive models will be developed utilizing genetic information obtained in Aim 1.1 and clinical data to predict treatment response
Development of a predictive model of leukemia toxicity | Day 28
  Predictive models will be developed utilizing genetic information obtained in Aim 1.1 and clinical data to predict treatment toxicity.

SECONDARY OUTCOMES:
Development of grade III/IV toxicity as defined by the CCG toxicity criteria | Day 28
  Contingency tables will be used to tabulate categorical toxicities and toxicity severity grade.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States